CLINICAL TRIAL: NCT02067676
Title: Safety and Immunogenicity Evaluation of an Intramuscular Capsule-Conjugate Campylobacter Vaccine (CJCV1)
Brief Title: Safety Study of a Capsule-Conjugate Vaccine to Prevent Campylobacter-Caused Diarrhea
Acronym: CJCV1-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-13-09; NMRC.2013.0021 (Other: Naval Medical Research Center IRB)
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Campylobacter Infection
Keywords: Campylobacter jejuni
MeSH Terms: conditions — Campylobacter Infections | interventions — Aluminum Hydroxide; aluminum sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CJCV1 2 μg / Alum 0 μg (1A) (Experimental): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 2 μg of polysaccharide and 0 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Interventions: Biological: Capsule-Conjugate Campylobacter Vaccine (CJCV1)
- CJCV1 2 μg / Alum 125 μg (1B) (Experimental): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 2 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Interventions: Biological: Capsule-Conjugate Campylobacter Vaccine (CJCV1); Drug: Alhydrogel®, aluminum hydroxide adjuvant (alum)
- CJCV1 5 μg / Alum 0 μg (2A) (Experimental): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 5 μg of polysaccharide and 0 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Interventions: Biological: Capsule-Conjugate Campylobacter Vaccine (CJCV1)
- CJCV1 5 μg / Alum 125 μg (2B) (Experimental): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 5 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Interventions: Biological: Capsule-Conjugate Campylobacter Vaccine (CJCV1); Drug: Alhydrogel®, aluminum hydroxide adjuvant (alum)
- CJCV1 10 μg / Alum 0 μg (3A) (Experimental): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 10 μg of polysaccharide and 0 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Interventions: Biological: Capsule-Conjugate Campylobacter Vaccine (CJCV1)
- CJCV1 10 μg / Alum 125 μg (1A) (Experimental): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 10 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Interventions: Biological: Capsule-Conjugate Campylobacter Vaccine (CJCV1); Drug: Alhydrogel®, aluminum hydroxide adjuvant (alum)

INTERVENTIONS:
Biological: Capsule-Conjugate Campylobacter Vaccine (CJCV1) — The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
Drug: Alhydrogel®, aluminum hydroxide adjuvant (alum)
  Arms: CJCV1 10 μg / Alum 125 μg (1A); CJCV1 2 μg / Alum 125 μg (1B); CJCV1 5 μg / Alum 125 μg (2B)

SUMMARY:
The purpose of this study is to assess the safety of increasing doses of a potential vaccine against Campylobacter with and without Alhydrogel®, an aluminum hydroxide adjuvant. This study will also assess immune responses induced by the vaccine.

DETAILED DESCRIPTION:
This is an open-label, dose-escalating study in which a total of 48 healthy volunteers will receive 2 vaccinations (one on Day 0 and one on Day 28 ± 2 days).

There are 3 cohorts (dose levels) with 2 groups of 8 volunteers in each cohort. A cohort will be administered one of 3 intramuscular (IM) doses at 2 μg, 5 μg, or 10 μg of Capsule-Conjugate Campylobacter Vaccine (CJCV1) with or without Alhydrogel®, aluminum hydroxide adjuvant (alum) at 125 μg.

An interval no less than 1 week will separate the last dose of a volunteer group from the first dose of the next volunteer group (receiving different CJCV1 doses). Blood specimens will be collected at intervals to examine systemic and mucosal antigen-specific immune responses. Vaccine safety will be actively monitored during vaccination and for 28 days (± 2 days) following the second vaccination and complete the study with a telephone follow-up approximately 6 months (± 1 month) after the first vaccination. The total duration of participation in this study is up to 270 days (including screening).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult, male or female, age 18 to 50 years (inclusive) at the time of enrollment.
* Completion and review of comprehension test (achieved 70% accuracy).
* Signed informed consent document.
* Available for the required follow-up period and scheduled clinic visits and telephone follow-up.
* Women: Negative pregnancy test with understanding (through informed consent) to not become pregnant during the study or within three months after the last vaccine dose (Day 28). Sexually active females, unless surgically sterile or at least one year postmenopausal, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device (IUD), female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner, or sterile sexual partner) prior to dosing of study vaccine. Female subjects unable to bear children must have a note from a primary care provider or obstetrics and gynaecology (OB/GYN) as proof of documentation (eg, tubal ligation or hysterectomy). If a volunteer becomes pregnant during the study, the PI will notify the study monitor, the sponsor, and the local institutional review board (IRB). The volunteer will be asked to provide serial follow-ups, including copies of clinic visits on the status of her pregnancy as well as health information on her infant following delivery.

Exclusion Criteria:

Health

1. Health problems affecting study participation from medical history (specifically to include chronic medical conditions such as diabetes mellitus and hypertension or any other condition requiring daily therapy that would place the volunteer at increased risk of adverse events (AEs). Study clinicians, in consultation with the PI, will use clinical judgment on a case-by-case basis to assess safety risks under this criterion. The PI will consult with the research monitor as appropriate.
2. Clinically significant abnormalities on physical examination
3. Use of immunosuppressive drugs, such as corticosteroids and chemotherapy, during the course of the study or immunosuppressive illness, including IgA deficiency (defined by serum IgA below level of detection)
4. Women who are pregnant or planning to become pregnant during the study period plus 3 months beyond the last vaccine dose and currently nursing women
5. Participation in research involving another investigational product 30 days before the planned date of first vaccination until the last study safety visit.
6. Positive blood test for HIV-1 (the human immunodeficiency virus and cause of AIDS)
7. Positive blood test for hepatitis B surface antigen (HBsAG; the virus causing hepatitis B)
8. Positive blood test for anti-HCV antibody (the virus causing hepatitis C)
9. Clinically significant abnormalities on basic laboratory screening
10. Presence of significant unexplained laboratory abnormalities that in the opinion of the PI may potentially confound the analysis of the study results Research Specific
11. Regular use (weekly or more often) of anti-diarrheal, anti-constipation, or antacid therapy
12. Abnormal bowel habits as defined by fewer than 3 stools per week or more than 3 loose/liquid stools per day
13. Personal or family history of inflammatory arthritis
14. Personal history of irritable bowel syndrome
15. Positive blood test for HLA-B27
16. History of allergy to any vaccine
17. History of allergy to alum
18. History of Guillain-Barré Syndrome or other neuroimmunological disorders Prior Exposure to Campylobacter
19. History of travelers' diarrhea or residence (> 2 months) in the past 3 years in a country with potentially higher Campylobacter rates to include Africa, South America, Central America, and Asia (except Japan).
20. Occupation involving handling of Campylobacter bacteria or vaccine products currently or in the past 3 years.
21. History of microbiologically confirmed Campylobacter infection.
22. Received previous experimental Campylobacter vaccine or live Campylobacter challenge.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2014-09-24 (Actual); Study Completion 2016-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro Gutierrez, MD, Principal Investigator — Enteric Disease Department, Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
WRAIR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 subjects participated at the Walter Reed Army Institute of Research (WRAIR), Clinical Trials Center (CTC).
Groups:
- CJCV1 2 μg / Alum 125 μg (1B): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 2 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Capsule-Conjugate Campylobacter Vaccine (CJCV1): The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
  Alhydrogel®, aluminum hydroxide adjuvant (alum)
- CJCV1 5 μg / Alum 125 μg (2B): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 5 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Capsule-Conjugate Campylobacter Vaccine (CJCV1): The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
  Alhydrogel®, aluminum hydroxide adjuvant (alum)
- CJCV1 10 μg / Alum 125 μg (1A): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 10 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  Capsule-Conjugate Campylobacter Vaccine (CJCV1): The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
  Alhydrogel®, aluminum hydroxide adjuvant (alum)
Period: Overall Study
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A)
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 8 | 8
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Customized [Count of Participants; unit: Participants]
  Age 18 to 50 years | 8 | 8 | 8 | 8 | 8 | 8 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 1 | 5 | 6 | 20
  Male | 6 | 6 | 4 | 7 | 3 | 2 | 28
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Safety: Presence of Related/Not Related Local and/or Systemic Reactogenicity (Adverse Events)
Description: Vaccine safety will be assessed by evaluating post-vaccination local and systemic reactions through targeted physical exams, symptom surveys, and other adverse event (AE) monitoring. All subjects will be observed in the clinic for at least 30 minutes after receipt of the investigational product. Approximately 48 hours after vaccination, subjects will return to the Clinical Trials Center for observation and reporting of any local and/or systemic AEs. Seven days after vaccine administration, subjects will return to the Clinical Trials Center to review their memory aids with study personnel and to report any AEs. In addition to planned visits, if a subject experiences any unanticipated AE, the subject will be seen by one of the study investigators. All AEs will be coded for onset date, duration, severity, and potential relationship to the investigational product.
Time Frame: up to 7 days
Population: Rates of all AEs were analyzed by Pearson's Chi-square test (or Fisher's exact test if assumptions were not met for Pearson's Chi-square) to compare groups.
Measure: Number; unit: Adverse Events
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Adverse Events
  AE's Related to Study Vaccine | 10 | 17 | 10 | 29 | 20 | 16
  Not Related to Study Vaccine | 12 | 22 | 8 | 3 | 20 | 9

2. Secondary Outcome: Frequency (%) of Vaccine-specific Immune Responses by Assay and Antigen Using Enzyme-linked Immunosorbent Assay (ELISA)
Description: Primary immunologic parameters, serum samples were assessed for the antibody titers against Campylobacter jejuni conjugate vaccine1 (CJCV1) using ELISA (enzyme-linked immunosorbent assay) based methods.
  Antibody-secreting cell(s) (ASCs): >0.5 per 10(6) Peripheral blood mononuclear cell (PBMCs) in the baseline sample. When the number of baseline ASCs is less than 0.5 per 10(6) PBMCs, a subject was considered a responder if the post-vaccination value was greater than 1.0 per 10(6) PBMCs. ((6) is superscript).
  1. = Seroconversion was defined as >4fold increase in endpoint titer between pre- and post-vaccine samples and a post-vaccine reciprocal titer >10.
  2. = Response is defined as a >2fold increase over the baseline value of ASC per 10(6) PBMCs, when the number of ASCs is >0.5 per 10(6) PBMCs in the baseline sample. When the number of baseline ASCs is less than 0.5 per 10(6) PBMCs, a subject was considered a responder if the post-vaccine value was greater than 1.0 per 10(6) PBMCs.
Time Frame: Study Days 0-56
Population: Campylobacter jejuni conjugate vaccine (1CJCV1); antibody-secreting cell(s) (ASCs); Peripheral blood mononuclear cell (PBMCs)
Measure: Number; unit: % of immune response
Groups:
- CJCV1 2 μg / Alum 0 μg (1A): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 2 μg of polysaccharide and 0 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  CJCV1: The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
- CJCV1 2 μg / Alum 125 μg (1B): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 2 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  CJCV1: The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
  Alhydrogel®, aluminum hydroxide adjuvant (alum)
- CJCV1 5 μg / Alum 0 μg (2A): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 5 μg of polysaccharide and 0 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  CJCV1: The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
- CJCV1 5 μg / Alum 125 μg (2B): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 5 μg of polysaccharide and 125 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum)
  CJCV1: The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
  Alhydrogel®, aluminum hydroxide adjuvant (alum)
- CJCV1 10 μg / Alum 0 μg (3A): Two vaccinations (one on Day 0 and one on Day 28) with an intramuscular dose of Capsule-Conjugate Campylobacter Vaccine (CJCV1) equivalent to 10 μg of polysaccharide and 0 μg of Alhydrogel®, aluminum hydroxide adjuvant (Alum) CJCV1: The capsule of Campylobacter jejuni strain 81-176 (CPS81-176) conjugated to the mutated diphtheria toxin cross-reacting material 197 (CRM197) (lyophilized CPS-CRM197 conjugate) (CJCV1)
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
% of immune response
  Serum IgG (CPS-BSA) (a) | 12.5 | 0 | 12.5 | 25.0 | 12.5 | 12.5
  Serum IgG (CRM197) (a) | 25.0 | 75.0 | 62.5 | 75.0 | 75.0 | 75.0
  IgG ASCs (CPS-BSA) (b) | 0 | 0 | 12.5 | 25.0 | 25.0 | 37.5
  IgG ASCs (CRM197) (b) | 87.5 | 100 | 87.5 | 100 | 100 | 87.5

3. Secondary Outcome: Vaccine-specific Geometric Mean Titers (GMT) of Anti-CPS IgG Antibody-secreting Cells
Description: Anti-CPS IgG ASC Responses - GMTs with 95% CI.
  A positive immunoglobulin A (IgA)-ASC response will be defined as a > twofold increase over the baseline value of the ASCs per 10^6 peripheral blood mononuclear cells (PBMCs). A subject will be considered a responder if the post-vaccination value is greater than 2.0 per 10^6 PBMCs. Blood samples will also be utilized to explore in vitro production of interferon (IFN)-(gamma).
Time Frame: Study Days 0-56
Measure: Geometric Mean (95% Confidence Interval); unit: GMTs
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
GMTs | 0 [0 to 0] | 1.1 [0.7 to 1.8] | 1.1 [0.6 to 2.2] | 1.9 [0.1 to 45.0] | 1.5 [0.4 to 5.9] | 1.3 [0.6 to 2.7]

4. Secondary Outcome: Vaccine-specific Anti-CRM^197 IgA Antibody-secreting Cell (ASC) Responses
Description: Anti-CRM^197 IgG ASC Responses - GMTs with 95% CI.
  A positive immunoglobulin A (IgA)-ASC response will be defined as a > twofold increase over the baseline value of the ASCs per 10^6 peripheral blood mononuclear cells (PBMCs). A subject will be considered a responder if the post-vaccination value is greater than 2.0 per 10^6 PBMCs. Blood samples will also be utilized to explore in vitro production of interferon (IFN)-(gamma).
Time Frame: Study Days 0-56
Measure: Geometric Mean (95% Confidence Interval); unit: GMTs
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
GMTs | 8.7 [0.2 to 308.3] | 16.0 [2.3 to 109.5] | 14.9 [0.8 to 272.3] | 35.3 [5.1 to 244.2] | 4.8 [0.9 to 24.7] | 10.2 [0.4 to 249.8]

5. Secondary Outcome: Interferon Titers Among All Cohorts
Description: CRM197-specific interferon-y (IFNy) responses measured from PBMC on day0, 28 and 56
Time Frame: Day 0, 28 and 56
Measure: Geometric Mean (95% Confidence Interval); unit: GMTs
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
GMTs | 44.3 [0.3 to 6920.3] | 45.5 [0.4 to 5657.0] | 154.9 [7.6 to 3174.0] | 195.4 [9.4 to 4076.3] | 153.5 [58.4 to 403.9] | 242.4 [37.1 to 1583.7]

ADVERSE EVENTS:
Time Frame: up to 7 days post-vaccination
Arm/Group | CJCV1 2 μg / Alum 0 μg (1A) | CJCV1 2 μg / Alum 125 μg (1B) | CJCV1 5 μg / Alum 0 μg (2A) | CJCV1 5 μg / Alum 125 μg (2B) | CJCV1 10 μg / Alum 0 μg (3A) | CJCV1 10 μg / Alum 125 μg (1A)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 8/8 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CJCV1 2 μg / Alum 0 μg (1A) (N=8) | CJCV1 2 μg / Alum 125 μg (1B) (N=8) | CJCV1 5 μg / Alum 0 μg (2A) (N=8) | CJCV1 5 μg / Alum 125 μg (2B) (N=8) | CJCV1 10 μg / Alum 0 μg (3A) (N=8) | CJCV1 10 μg / Alum 125 μg (1A) (N=8)
Acute pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CJCV1 2 μg / Alum 0 μg (1A) (N=8) | CJCV1 2 μg / Alum 125 μg (1B) (N=8) | CJCV1 5 μg / Alum 0 μg (2A) (N=8) | CJCV1 5 μg / Alum 125 μg (2B) (N=8) | CJCV1 10 μg / Alum 0 μg (3A) (N=8) | CJCV1 10 μg / Alum 125 μg (1A) (N=8)
Adbominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Related
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Related
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Related
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Related
Loose stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Related
LUE pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Related
LUE tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Related
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Related
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Related
Phantom sensation LUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Related
Sweats (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related
Vaccine site ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Related
Vaccine site erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 4 (4) | 2 (2) — Related
Vaccine site induration (General disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 2 (2) — Related
Vaccine site nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Related
Vaccine site pain (General disorders) | 2 (2) | 3 (3) | 1 (1) | 6 (6) | 1 (1) | 1 (1) — Related
Vaccine site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Related
Vaccine site tenderness (General disorders) | 3 (3) | 6 (6) | 2 (2) | 8 (8) | 7 (7) | 8 (8) — Related
Abdominal pain/cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Unrelated
Acute pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Allergic rhinitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated
Allergy headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Ankel sprain-right (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Decreased blood glucose (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Decreased platelets (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Ecchymosis LUE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Elevated ALT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Elevated AST (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Elevated blood glucose (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Elevated cosinophils (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Elevated WBC (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Feverish chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Gastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Hangover symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Unrelated
Hemoglobin decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Unrelated
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Increased cosinophil (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Left eyelid twitching (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated
Loose stool (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Unrelated
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — Unrelated
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — Unrelated
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Unrelated
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Right fingertip pareshesias (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Soft tissue chest muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Sweats (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Unrelated
Upper respiratory infection symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No